CLINICAL TRIAL: NCT06878001
Title: CaroRite™ for Improving Skin Health and the Visible Signs of Ageing, a Placebo Controlled, Double Blind, Randomised Clinical Trial
Brief Title: CaroRite™ for Skin Health and Signs of Ageing
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: RDC Clinical Pty Ltd (Industry)
Collaborators: Bio-Gen Extracts Pvt. Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIOCAR
Record Dates: First submitted 2025-03-04; First posted 2025-03-14 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-03

CONDITIONS: Healthy Volunteer; Skin Condition; Ageing Signs
Keywords: females; Skin Health; Carotenoids
MeSH Terms: conditions — Skin Diseases | interventions — Carotenoids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CaroRite (Experimental): CaroRite capsule containing carotenoids with sunflower oil. 1 capsule to be taken each day for 12 weeks.
  Interventions: Dietary Supplement: Carotenoids
- Placebo (Placebo Comparator): Placebo capsule containing sunflower oil. 1 capsule to be taken each day for 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Carotenoids — CaroRite capsule containing carotenoids with sunflower oil. 1 capsule to be taken each day for 12 weeks.
  Other Names: CaroRite
  Arms: CaroRite
Other: Placebo — Placebo capsule containing sunflower oil. 1 capsule to be taken each day for 12 weeks.
  Arms: Placebo

SUMMARY:
The goal of this study is to investigate the efficacy of carotenoids administered orally on skin health, skin condition and visible signs of ageing in healthy females aged 40-55 years old.

Researchers will compare the study product against placebo.

ELIGIBILITY:
Inclusion Criteria:

* Females 40-55 years (inclusive)
* Generally healthy
* BMI 18.5-29.9 kg/m2 (inclusive)
* Able to provide informed consent
* Agree not to change regular skincare routine
* Agree to not participate in another clinical trial while enrolled in this trial
* Agree to not significantly change current diet and/or exercise frequency or intensity during study period

Exclusion Criteria:

* Regularly taking carotenoid containing medication/supplements within the previous 2 months
* Have a serious illness e.g. mood disorders such as clinical depression, anxiety disorder or bipolar disorder, neurological disorders such as MS, kidney disease, liver disease or heart conditions
* Have an unstable illness e.g. diabetes and thyroid gland dysfunction
* Current malignancy (excluding Basal Cell Carcinoma) or chemotherapy or radiotherapy treatment for malignancy within the previous 2 years
* Received cosmetic surgery or procedures, including Botox and other injectables, microdermabrasion and laser treatments on their face within last 3 months prior to enrolment and agree not to have these treatments during the study period.

  * Medications for acne or other skin conditions including topical retinoids (Rein-A, Retrieve) oral retinoids such as Isotretinoin (Roaccutane), benzoyl peroxide, AHA's, serum, chemical peels within 1 month prior to screening.
  * Currently taking carotenoid supplements (Beta-Carotene, Lycopene, Lutein, Zeaxanthin, Astazanthin)
  * Active smokers, nicotine use or drug (prescription or illegal substances) abuse
  * Chronic past and/or current alcohol use (>14 alcoholic drinks week)
  * Pregnant or lactating women
  * Allergic to any of the ingredients in active or placebo formula
  * Participants who are currently participating in any other clinical trial or who have participated in a clinical trial that may affect skin health during the past 1 month
  * Any condition which in the opinion of the investigator makes the participant unsuitable for inclusion

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to the end of the study period in Visible signs of ageing | Baseline to week 12
  Assessed using the A-One Smart Pro, this device provides and automatic skin analysis by scanner and multi-sensor. It uses a high-resolution camera to take photographs of the skin in normal, UV and polarized light. Wrinkles will be measured as thin and thick and rated on a scale of 1-10 in each area of the face: forehead, eyes, mouth and nose. An attached probe measures skin temperature and moisture.
  Visible signs of ageing measured include:
  * Skin elasticity
  * Hydration
  * Wrinkle depth and type
  * Sebum
  * pigmentation
  * Skin pH and temperature

SECONDARY OUTCOMES:
Change from baseline to the end of the study period in Transepidermal water loss (TEWL) | Baseline to week 12
  Change from baseline to the end of the study period in Transepidermal water loss (TEWL). Analysed using a DermaLab Combo system with a probe for measurement.
Change from baseline to the end of the study period in Skin collagen thickness | Baseline to week 12
  Change from baseline to the end of the study period in Skin collagen thickness. Analysed using the DermaLab Combo system with a probe to measure.
Change from baseline to the end of the study period in Skin carotenoid analysis | Baseline to week 12
  Change from baseline to the end of the study period in Skin carotenoid analysis. This will be measured using a non-invasive device that measures skin carotenoid levels using reflection spectroscopy.
Change from baseline to the end of the study period in Safety and adverse events | Baseline to week 12
  Change from baseline to the end of the study period in Safety and adverse events. At each point of contact the participant will be asked about adverse events they may have experienced.
Change from baseline to the end of the study period in Participant self-assessment of product effectiveness | Baseline to week 12
  Change from baseline to the end of the study period in Participant self-assessment of product effectiveness. This Consists of questions related to overall satisfaction with the product and specific facial and skin properties
Change from baseline to the end of the study period in Self-administered carotenoid intake questionnaire | Baseline to week 12
  Change from baseline to the end of the study period in Self-administered carotenoid intake questionnaire. The questionnaire consists of 17 questions related to overall satisfaction with the product and specific facial and skin properties.
Change from baseline to the end of the study period in 24-hour diet recall | Baseline to week 12
  Change from baseline to the end of the study period in 24-hour diet recall
Skin carotenoid analysis (Veggie Metre) | Baseline to week 12
  Change from baseline to the end of the study period in Skin carotenoid analysis (Veggie Metre). Analysed using the Veggie Meter analyser. The Veggie Meter® is a non-invasive device that measures skin carotenoid levels using reflection spectroscopy. It shines a specific wavelength of light onto the skin (typically from an LED) and analyses the light that is absorbed and reflected. Carotenoids absorb certain wavelengths of light, and the device quantifies this absorption to determine carotenoid concentration in the skin.

CONTACTS AND LOCATIONS:
Overall Officials: Salman Mehkri, Study Director — Bio-gen Extracts
Locations (1):
- RDC Clinical, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: Undecided